CLINICAL TRIAL: NCT03487185
Title: A Randomized Trial of Continuous Positive Airway Pressure (CPAP) for Sleep Apnea in Pregnancy
Brief Title: Continuous Positive Airway Pressure (CPAP) for Sleep Apnea in Pregnancy
Acronym: SLEEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HD36801-SLEEP; U24HD036801 (NIH); UG1HD087192 (NIH); UG1HD087230 (NIH); UG1HD027869 (NIH); UG1HD034208 (NIH); UG1HD053097 (NIH); UG1HD040500 (NIH); UG1HD040485 (NIH); UG1HD040544 (NIH); UG1HD040545 (NIH); UG1HD040560 (NIH); UG1HD040512 (NIH); UG1HD027915 (NIH); UG1HD112096 (NIH); UG1HD112063 (NIH); UG1HD112092 (NIH)
Record Dates: First submitted 2018-03-22; First posted 2018-04-03 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea of Adult; Preeclampsia; Obstetrical Complications
Keywords: CPAP; Apnea; pregnancy
MeSH Terms: conditions — Pre-Eclampsia; Apnea | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Women who are between 14 weeks 0 days and 21 weeks 5 days with a singleton gestation and obstructive sleep apnea (OSA) will be randomized to one of two arms at participating MFMU Network clinical center:
  * Autotitrating CPAP with weekly contact, incentives for compliance and initial sleep advice counseling
  * Initial sleep advice counseling alone
Who Masked: Investigator, Outcomes Assessor
Masking Description: This study is an unmasked randomized controlled multi-center clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Continuous Positive Airway Pressure (Experimental): Autotitrating CPAP with weekly contact, incentives for compliance and initial sleep advice counseling
  Interventions: Device: Continuous Positive Airway Pressure
- Sleep Advice Control (Other): Initial sleep advice counseling alone
  Interventions: Other: Sleep Advice Control

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — Autotitrating CPAP with weekly contact, incentives for compliance and initial sleep advice counseling
  Other Names: CPAP
  Arms: Continuous Positive Airway Pressure
Other: Sleep Advice Control — Initial sleep advice counseling alone
  Arms: Sleep Advice Control

SUMMARY:
A randomized controlled trial of 1,500 women to assess whether treatment of obstructive sleep apnea with continuous positive airway pressure (CPAP) in pregnancy will result in a reduction in the rate of hypertensive disorders of pregnancy.

DETAILED DESCRIPTION:
Emerging data support a link between sleep disordered breathing (SDB) and adverse pregnancy outcomes. In particular, women with obstructive sleep apnea (OSA) appear to be at increased risk of both hypertensive disorders of pregnancy and gestational diabetes. In the non-pregnant population, OSA is typically treated with continuous positive airway pressure (CPAP) during sleep and has been shown to reduce blood pressure in hypertensive patients. Unfortunately, data on whether maternal and neonatal outcomes could be improved with treatment of OSA during pregnancy are extremely limited. This study aims to address this knowledge gap.

A randomized controlled trial of 1,500 women to assess whether treatment of obstructive sleep apnea with continuous positive airway pressure (CPAP) in pregnancy will result in a reduction in the rate of hypertensive disorders of pregnancy.

ELIGIBILITY:
Inclusion Criteria

1. Singleton gestation. Twin gestation reduced to singleton, either spontaneously or therapeutically, is not eligible unless the reduction occurred before 14 weeks project gestational age.
2. Gestational age at randomization between 14 weeks 0 days and 21 weeks 6 days based on clinical information and evaluation of the earliest ultrasound.
3. Diagnosis with mild to moderate OSA as defined by an AHI score ≥ 5 and <30.

Exclusion Criteria

1. Previously prescribed, current or planned therapy for sleep apnea.
2. Age < 18 years, because the rate of sleep apnea in this population is extremely low.
3. Inability to sleep in a stable place with access to the CPAP machine at least 5 nights per week.
4. Asthma requiring systemic steroid therapy for more than 14 days within the past 6 months because this population is expected to be unresponsive to CPAP therapy.
5. Current use of prescribed sleeping pills for insomnia.
6. Chronic medical conditions requiring oxygen supplementation (e.g. pulmonary fibrosis, pulmonary hypertension, cystic fibrosis) because this population is expected to be unresponsive to CPAP therapy.
7. Chronic renal disease with serum creatinine >1.3 mg/dL because the primary outcome would be pre-determined.
8. Antiphospholipid antibody syndrome, because it would compromise the primary outcome diagnosis.
9. History of medical complications such as:

   1. Active liver disease (acute hepatitis, chronic active hepatitis, persistently abnormal liver enzymes)
   2. Thrombocytopenia with platelet count <100,000 because of the difficulty in assessing the primary outcome.
10. Active vaginal bleeding (more than spotting) at the time of randomization.
11. Known chromosomal, genetic, major malformations or fetal demise, or planned termination of pregnancy because inclusion would compromise evaluation of secondary neonatal outcomes.
12. Known major uterine malformations associated with adverse pregnancy outcomes.
13. Current use of opiates (heroin, methadone, or other daily opioid use) due to inaccuracy of the home sleep test and inefficiency of CPAP.
14. Active drug use, alcohol use, or unstable psychiatric condition.
15. Participation in another interventional study that influences preeclampsia, hypertensive disorders of pregnancy, or GDM.
16. Prenatal care or delivery planned at a non-network center where access to the complete electronic medical record will not be available to research staff.
17. Participation in this trial in a previous pregnancy. Patients who were screened in a previous pregnancy, but not randomized, may be included.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2018-08-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Hypertensive Disorders of Pregnancy | Up to 14 days postpartum
  Subjects are considered to have the primary outcome if they meet the criteria for eclampsia, HELLP, atypical HELLP, preeclampsia, superimposed preeclampsia or antepartum gestational hypertension.

SECONDARY OUTCOMES:
Gestational diabetes | As soon as possible after randomization between 14 weeks, 0 days and 21 weeks, 6 days gestation
  Gestational diabetes by oral GTT criteria performed after randomization
Preterm birth | Preterm delivery up to and less than 37 weeks gestation
  Preterm birth less than 34 weeks and less than 37 weeks
Cesarean Delivery | At the time of delivery
  Delivery by cesarean section
Maternal morbidity composite | Within 6 weeks postpartum
  Maternal morbidity composite defined as the occurrence of one of the following:
  * Maternal death
  * Transfusion of ≥ 4 units of PRBC within 6 weeks postpartum
  * ICU admission within 6 weeks postpartum
Maternal adverse cardiovascular outcome composite | By 6 weeks postpartum
  Maternal adverse cardiovascular outcome composite defined as the occurrence of one or more of the following:
  * Venous thromboembolism
  * New onset heart failure with ejection fraction (EF) < 40%
  * Cerebrovascular accident
  * Myocardial infarction
  * New onset atrial fibrillation
Fetal or Neonatal Death | through 72 hours postpartum
  Antepartum, intrapartum, or neonatal death
Neonatal respiratory support | within 72 hours of delivery
  Intubation, continuous positive airway pressure (CPAP) or high-flow nasal cannula (HFNC) for ventilation or cardiopulmonary resuscitation
Birth weight | Immediately post birth
  1. Small for gestational age defined as < 5th percentile weight for gestational age, assessed specifically by sex and race of the infant based on United States birth certificate data
  2. Large for gestational age defined as greater than the 90th percentile for gestational age.
  3. Macrosomia defined as birthweight > 4000 grams
Neonatal encephalopathy | within 72 hours of delivery
  Neonatal encephalopathy as defined by the NICHD Neonatal Research Network criteria
Neonatal Seizures | 72 hours post birth
  Neonatal seizure activity confirmed by central review
Shoulder dystocia | During delivery
  Shoulder dystocia during delivery
Birth trauma | During delivery
  Bone fractures, brachial plexus palsy, other neurologic injury, retinal hemorrhage, or facial nerve palsy
Intracranial hemorrhage | Within 72 hours post delivery
  Intraventricular hemorrhage grades III and IV, subgaleal hematoma, subdural hematoma, or subarachnoid hematoma
Hyperbilirubinemia | Within 72 hours post delivery
  Hyperbilirubinemia requiring phototherapy or exchange transfusion
Hypoglycemia | Within 72 hours post delivery
  glucose < 35 mg/dl requiring IV therapy
NICU Stay | Greater than or equal to 72 hours post birth
  Neonatal Intensive Care Unit stay

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Clifton, PhD, Principal Investigator — The George Washington University Biostatistics Center; Monica Longo, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Francesca Facco, MD, Study Chair — Magee Women's Hospital of UPMC
Locations (14):
- United States (14):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Regents of the University of California San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Case Western Reserve-Metro Health, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - Brown Univeristy, Providence, Rhode Island
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be shared per NIH policy after the completion and publication of the main analyses.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Facco F. Sleep Duration, Sleep Timing, and Sleep Disordered Breathing-Associations With Obesity and Gestational Diabetes in Pregnancy. Clin Obstet Gynecol. 2021 Mar 1;64(1):196-203. doi: 10.1097/GRF.0000000000000587. PMID 33481418